CLINICAL TRIAL: NCT04378673
Title: Pediatric Nursing in Bagcilar Training and Research Hospital
Brief Title: The Effect of Parental Presence on Pain and Anxiety Levels During Peripheral Intravenous Catheterization in Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16867222; Seda Caglar (Other: Istanbul University Cerrahpaşa)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Family Centered Care
Keywords: family centered care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- parental involvement group: n=46
- parental presence group: n=42
- parental absence group: control group, n=32
  Interventions: Other: not interventional

INTERVENTIONS:
Other: not interventional — This randomized controlled trial included data from 120 cases in the pediatric health and diseases department.
  Groups: parental absence group

SUMMARY:
Children's changing emotional and physical needs, continuous, comprehensive, accessible, coordinated and family requires a centered care.Parental presence during invasive procedures is important in family-centered-care. Family-centered-care is a basic principle of pediatric nursing. It is extremely important that parents are with their children during painful procedures. Research; parents during peripheral intravenous catheterization in infancy It was planned to determine the effect of inclusion on pain and anxiety.

DETAILED DESCRIPTION:
This randomized controlled trial included data from 120 cases in the Pediatric Health and Diseases Department of Istanbul, during March 2020-August 2020 (parental involvement group, n = 46; parental presence group, n = 42; parental absence group, n = 32). Information form, State-Trait Anxiety Inventory and FLACC scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Children within the age group of 1-24 months Parents know Turkish language

Exclusion Criteria:

-

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants and their parents were randomly sampled from the universe using a simple random sampling method, peripheral intravenous catheterization, volunteering to participate in the study, infants and parents between 1 and 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
hypothesis 0 | March 2020-August 2020
  There is no difference between the pain and anxiety levels of the children whose parents were included in the procedure during peripheral intravenous catheterization and the pain and anxiety levels of the children whose parents were only with the child during the procedure and who were not with the child during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Demir, Nurse, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training And Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided